CLINICAL TRIAL: NCT06495684
Title: Effects of Multiple-Session Transcranial Direct Current Stimulation (tDCS) on Behavioral, Physiological, and Electrophysiological Measures With Adults With Autism Spectrum Disorder (ASD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 24-059; P20GM109089 (NIH)
Record Dates: First submitted 2024-06-25; First posted 2024-07-11 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder; Autism or Autistic Traits
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Within-subject, cross-over, double-blind, randomized controlled trial
Who Masked: Participant, Investigator
Masking Description: Participants will receive 5 sessions of active tDCS in one block and 5 sessions of sham tDCS in another block. The tDCS device allows for researchers and participants to remain blind to the condition until the end of the study by randomly assigning participants to either the active or the sham block and providing the study team members a unique code to enter into the tDCS device at the start of each session.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Anodal tDCS + Social Learning (Experimental): In this arm, participants will undergo 5 sessions of 30 minutes anodal tDCS combined with social learning tasks on consecutive weekdays.
  Interventions: Device: Anodal tDCS + Social Learning
- Placebo anodal tDCS + Social Learning (Sham Comparator): In this arm, participants will undergo 5 sessions of 30 minutes placebo anodal tDCS combined with social learning tasks on consecutive weekdays.
  Interventions: Behavioral: Placebo Anodal tDCS + Social Learning

INTERVENTIONS:
Device: Anodal tDCS + Social Learning — Anodal tDCS lowers neuronal membrane potentials, leading to increased probability of depolarization from incoming stimuli.
  Arms: Anodal tDCS + Social Learning
Behavioral: Placebo Anodal tDCS + Social Learning — Social learning tasks are completed on a computer and consist of viewing video modeling of social interactions, facial emotion detection practice, and videos for emotion and empathy learning.
  Arms: Placebo anodal tDCS + Social Learning

SUMMARY:
The purpose of this clinical trial is to investigate the effects of multiple sessions of transcranial direct current stimulation (tDCS) delivered while participants complete tasks that target social learning with high functioning adults with ASD and/or high traits of ASD.

The main question it aims to answer is:

What are the effects of multiple sessions of active compared to sham tDCS, with tDCS simultaneously paired with social learning tasks, from employing a within-subject, cross-over randomized controlled trial design?

Participants will:

* Complete a randomly assigned block of 5 sessions of active and a block of 5 sessions of sham tDCS, with a four-week break occurring between the two blocks.
* Complete social learning tasks simultaneously during receipt of tDCS at each session (whether receiving active or sham tDCS).
* Complete behavioral, physiological, and electrophysiological testing before and after each block of active or sham tDCS.
* Complete a social validity questionnaire after completion of the study.

DETAILED DESCRIPTION:
Our long-term goal is to develop safe and effective treatments to reduce negative symptoms of social communication impairments to improve overall quality of life. Our central hypotheses are (1) active, anodal tDCS over the right temporoparietal junction (rTPJ) paired with social learning activities will result in improved performance on behavioral and physiological measures, when compared to sham stimulation, (2) these improvements in performance will be correlated with changes in electrophysiological measures that contribute to successful participant social alignment after receipt of anodal tDCS, such as reductions in spectral alpha power (8-12Hz), which has been robustly associated with accurate internal modeling of sensorimotor activity during action comprehension and speech perception, and (3) improvements in performance on social measures will be accompanied by power reductions in theta oscillations (4-8Hz), which arise from prefrontal cortices and support context-specific cognitive control.

Specific Aim 1: Determine the effects of multiple sessions of active compared to sham tDCS. This aim will employ a within-subject, cross-over randomized controlled trial (RCT) design to explore the effects of 5 sessions of active vs. 5 sessions of sham tDCS on behavioral, physiological, and electrophysiological measures with autistic adults or adults with high traits of autism.

Objective 1: The development of improved stimulation protocols

While even a single session of tDCS has been shown to improve performance on social measures with adults diagnosed with autism spectrum disorder (ASD), recent work with children with ASD has shown that increasing the number of sessions from one to even five produces positive effects that are retained for up to one year, even when tDCS was not paired with a task. Importantly, it has been shown that pairing a task with the receipt of tDCS improves results when compared to delivering tDCS without a task. However, the majority of literature on the use of tDCS with adults with ASD has been restricted to studies examining a low number of sessions and/or tDCS paired with no task or tasks that are unrelated to treating the core diagnostic social impairments of ASD. This reinforces the need for research examining multiple sessions of tDCS paired with social interventions that are relevant to core diagnostic social impairments in autistic adults or adults with high traits of autism.

Objective 2: The improvement of social communication and social alignment in autistic adults or adults with high traits of autism

Successful social communication is a complex social process that not only requires the expression and reception of verbal speech, but also the modification and coordination of many behaviors to achieve social alignment. Social alignment is a mostly unconscious phenomenon in which people become more similar to a conversation partner by adjusting communication features such as vocal speech prosody (patterns of voice stress or intonation), facial expressions, and gestures.It is also suggested that social alignment reduces the burden placed on the cognitive system, thus making social interactions easier, and possibly less anxiety filled. Autistic individuals have significantly lower social alignment when compared to their neurotypical peers.

Of great interest is also capitalizing on the rTPJ's role in social alignment because of the rTPJ's participation in using sensory information (including visual and auditory) to evaluate self against others and in mediating embodied processes relevant to perspective taking (such as facial expression and gesture). Consequently, the proposed project has significance in its approach for investigating tDCS applied over the rTPJ that is paired with social learning to target processes of social communication and social alignment in autistic adults or adults with high traits of autism.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-35 years
2. Proficient in English
3. Classification of autism or autism spectrum disorder on Autism Diagnostic Observation Scale, 2nd Edition (ADOS-2) or score of >= 17 on Autism Quotient (AQ)
4. Good or corrected vision and hearing
5. Right-handed based on the Edinburgh Handedness Inventory
6. Score of >= 85 on Shipley-2

Exclusion Criteria

1. No known loss of consciousness for > 5 minutes
2. No immediate biological family members with a history of epilepsy or seizure disorder
3. No major medical needs (e.g., neurological disorders such as a seizure disorder; long-term illness)
4. No surgically implanted metal above the neck (example: metal pins or plates, cochlear implants, aneurysm clips, brain electrodes)
5. No hospitalization for depression, anxiety, or substance abuse in the past 12 months
6. No individuals who are currently pregnant
7. No pacemakers
8. No history of neurological disorders such as stroke, multiple sclerosis, bipolar disorder, encephalitis, epilepsy, seizure disorder, or amyotrophic lateral sclerosis

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Measure of Emotional Distress - Anxiety | Before and after each 5-day block of tDCS stimulation
  Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v. 1.0 - Emotional Distress - Anxiety (PEDA) A change in PEDA scores corresponds to a change in emotional distress and anxiety. Each question on the PEDA provides a 5-point scale where lower scores mean a better outcome.
Measure of Social Anxiety | Before and after each 5-day block of tDCS stimulation
  Liebowitz Social Anxiety Scale (LSAS) The LSAS assesses the range of social interaction and performance situations that individuals with social anxiety may fear and/or avoid. Each two-part question of the LSAS provides a 4-point scale where lower scores mean a better outcome.
Measure of Social Anxiety/Anxiety | Before and after each 5-day block of tDCS stimulation
  Vocal acoustic analysis measures changes in fundamental frequency (F0), which is an indicator of change in social anxiety/anxiety, where lower F0 means a better outcome.
Measure of Social Anxiety | Before and after each 5-day block of tDCS stimulation
  Heart-Rate Variability (HRV) A change in HRV is an indicator of change in the level of social anxiety, where higher HRV means a better outcome.
Measure of Social Impairment | Before and after each 5-day block of tDCS stimulation
  Social Responsiveness Scale - 2nd Edition (SRS-2) A self-report tool that quantifies social impairment and its severity associated with ASD. Lower SRS-2 scores mean a better outcome.
Measure of Empathy | Before and after each 5-day block of tDCS stimulation
  Empathy Quotient (EQ) A self-report measure that quantifies empathy. Higher EQ scores mean a better outcome.
Measure of Prosodic Alignment | Before and after each 5-day block of tDCS stimulation
  Vocal acoustic analysis measures the rate of prosodic alignment between speakers sharing in a conversation. Higher rates of prosodic alignment between speakers mean a better outcome.
Measure of Emotion Expression Entrainment | Before and after each 5-day block of tDCS stimulation
  Facial expression and gesture analysis measures the rate of emotion entrainment to others during conversation tasks. Increased rate of emotion entrainment means a better outcome.
Measure of Social Learning | Before and after each 5-day block of tDCS stimulation
  Electroencephalography (EEG) spectral power for alpha (8-12Hz) and theta (4-8Hz) oscillations measures changes in social learning. Reductions in power for alpha and theta mean a better outcome.
Measure of Quality of Life | Before and after each 5-day block of tDCS stimulation
  World Health Organization Quality of Life Questionnaire (WHOQOL) The WHOQOL measures quality of life in areas of social relationships, psychological and physical health, environment, and independence. Higher WHOQOL mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Bill Shuttleworth, Ph.D., Study Director — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States